CLINICAL TRIAL: NCT03423927
Title: Benefits of an Intervention Combining Hypnosis and Self-care for Prostate Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: Free University of Brussels (Other)
Responsible Party: Principal Investigator, Isabelle Bragard, Lecturer, University of Liege
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Hypnosis Prostate Cancer
Record Dates: First submitted 2018-01-30; First posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Hypnosis; Self Care

STUDY DESIGN:
Intervention Model Description: Participants who agree to participate in the intervention are assigned in the experimental group, whereas participants who do not agree to participate in the intervention, but agree to answer the questionnaires, are assigned in the control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group : hypnosis + self-care (Experimental): Groupal intervention combining self-care techniques and self-hypnosis exercises
  Interventions: Behavioral: Self-hypnosis + Self-care
- Control group : no intervention (No Intervention): Control group receiving usual care but not the intervention

INTERVENTIONS:
Behavioral: Self-hypnosis + Self-care — Our groupal intervention is divided into 6 monthly 2-hour sessions in which one self-hypnosis exercise is proposed to participants. Self-care techniques are also discussed (knowing our own needs, selfrespect, assertiveness, coping with ruminations...) and homework assignments are proposed to participants, in order to foster positive change.
  Arms: Intervention group : hypnosis + self-care

SUMMARY:
This study aims to assess the impact of a group intervention combining self-hypnosis and self-care techniques on prostate patients' well-being. More specifically, the investigators want to investigate the effects of that intervention on sleep, fatigue and emotional distress of the patients.

ELIGIBILITY:
Inclusion Criteria:

* 18-years-old,
* ability to read, write and speak French
* prostate cancer diagnosis
* treatment with surgery and/or radiotherapy.

Exclusion Criteria:

* metastases
* cancer recurrence at the moment of inclusion
* major cognitive or psychiatric disorder.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-10-14 (Actual); Primary Completion 2016-06-15 (Actual); Study Completion 2016-06-15 (Actual)

PRIMARY OUTCOMES:
Change in Fatigue | T0 (before the intervention) and T1 (after the intervention : 6 months later).
  A sense of tiredness or exhaustion linked with cancer and its treatments, that is not alleviated by sleep. Measured by the European Organization for Research and Treatment of Cancer - Quality of Life Core Questionnaire-30 (EORTC-QLCQ30). One symptom-related scale (fatigue, score based on 3 items, varies from 0 to 100, 100 being the worst fatigue endured) and the global health status (2 items, score varies from 0 to 100, 100 being the best quality of life) are used in this study.
Change in emotional distress | T0 (before the intervention) and T1 (after the intervention : 6 months later).
  Anxiety + Depression, measured with the Hospital Anxiety and Depression Scale (HADS). Scores range (total): 0-42 (0-14: absence of anxio-depressive disorder ; 15-42: presence of anxio-depressive disorder). Two scales: anxiety and depression. For each, scores range 0-21 (0-7: absence of anxious or depressive disorder; 8-10: possibility of an anxious or depressive disorder; 11-21: presence of anxious or depressive disorder).
Change in sleep difficulties | T0 (before the intervention) and T1 (after the intervention : 6 months later).
  Sleep difficulties (difficulties to stay asleep, to fall asleep...) and their severity. Measured by the Insomnia Severity Index. One score is calculated and ranges from 0 to 22 (0-7: absence of insomnia; 8-14: subclinical insomnia; 15-21: moderate insomnia; 22-28: severe insomnia).

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Elisabeth Faymonville, Study Director — University of Liege

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gregoire C, Nicolas H, Bragard I, Delevallez F, Merckaert I, Razavi D, Waltregny D, Faymonville ME, Vanhaudenhuyse A. Efficacy of a hypnosis-based intervention to improve well-being during cancer: a comparison between prostate and breast cancer patients. BMC Cancer. 2018 Jun 22;18(1):677. doi: 10.1186/s12885-018-4607-z. PMID 29929493